CLINICAL TRIAL: NCT00938496
Title: A Non-interventional Study of Postoperative Treatment With Goserelin Acetate (Zoladex) in Moderate to Severe Endometriosis Patient
Brief Title: Non-Interventional Study of Zoladex in Endometriosis
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-ZOL-2009/1
Record Dates: First submitted 2009-07-09; First posted 2009-07-14 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, open label NIS, which is to assess the efficacy of Zoladex in adjuvant setting after operation in moderate to severe endometriosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced endometriosis confirmed histologically (r-AFS score III-IV) with conservative laparoscopy or laparotomy.
* Patient who has the indication of Zoladex and has been prescribed Zoladex according to physician's judgement, irrespective of the inclusion in the study.
* Patient has been already prescribed Zoladex within 1 month after operation.

Exclusion Criteria:

* Have used hormone treatment prior to 3 months of recruitment.
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site).
* Previous enrolment in the present study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description: Patient with advanced endometriosis confirmed histological (r-AFS score III-IV) with conservative laparoscopy or laparotomy has the indication of Zoladex and has already been prescribed Zoladex according to physician's judgment, irrespective of the inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Symptom recurrence rate and total recurrence rate | 18 months

SECONDARY OUTCOMES:
Pregnancy rate | 18 months
Zoladex administration time | 6 months
Add-back therapy information | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Yingfang, Principal Investigator — Peking University First Hospital
Locations (11):
- China (11):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Changsha, Hunan
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- See also: CSR-NIS-OCN-ZOL-2009-1.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=980&filename=CSR-NIS-OCN-ZOL-2009-1.pdf